CLINICAL TRIAL: NCT03967769
Title: Apneic Oxygénation by Nasal Canula During Infants Airway Management Study
Acronym: Oxyeno
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Oxyneo; 2018-004127-36 (EudraCT Number)
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Infant Apnea; Surgical Procedure, Unspecified; Airway Management
Keywords: Apnoeic oxygenation; Airway management; Oxygen insufflation; Paediatric general anaesthesia

STUDY DESIGN:
Intervention Model Description: Monocentric prospective, randomized, stratified, parallel-group clinical trial with concealed allocation to 3 groups of Apnoeic Oxygenation during Airway management for general anesthesia in elective surgery.
  All participants will receive French actual standard of care of surgery and anesthesia.
Who Masked: Participant, Care Provider, Investigator
Masking Description: At each participating center, patients will be followed up for primary and secondary endpoints by members of the research staff who will be unaware of the trial group allocation. Information on whether the primary and secondary outcomes occur will be collected and entered into the electronic web-based case report form (eCRF) by trial or clinical trained personal (clinical research associate), blinded to the allocation group, under the supervision of the local principal investigator (PI) or designee who will also be unaware of the trial group allocation.
  Finally, the independent trial statistician and the members of the data monitoring and safety committee (DMSC) will also remain blinded for the allocation during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Practice (No Intervention): Infants will have high Flow nasal cannulae placed into the nares before induction. They will be removed from the nares at the end of the study when the airway has been secured. There will be no oxygen flowing through the cannulae in this group during the study.
- Low Flow oxygenation (Experimental): Infants will have conventional nasal cannulae into the nares prior to induction of anesthesia. They will be removed from the nares at the end of the study when the airway has been secured. There will be 0,2L/kg/min of oxygen flowing through the cannulae in this group during the study.
  Interventions: Device: High Flow nasal Cannula
- High Flow Oxygenation (Experimental): Infants will have conventional nasal cannulae into the nares prior to induction of anesthesia. They will be removed from the nares at the end of the study when the airway has been secured. There will be 1L/kg/min of oxygen flowing through the cannulae in this group during the study.
  Interventions: Device: High Flow nasal Cannula

INTERVENTIONS:
Device: High Flow nasal Cannula — Apnoeic Oxygenation by High Flow Nasal Cannulae
  Arms: High Flow Oxygenation; Low Flow oxygenation

SUMMARY:
This is a randomized clinical trial investigating the utility of apneic oxygenation via high flow nasal cannulae during airway management for infants general anaesthesia. Three groups will be compared, a control group at 0 L/min, a 0,2L/Kg/min and a 1L/Kg/min group. The primary outcome will be the time (in seconds) between onset of apnea and one of theses end-points : desaturation (SPO2 <95%) or Airway management completed.

DETAILED DESCRIPTION:
Airway management can be a life saving therapy. One major complication that may occur during airway management is a lack of oxygen in the blood, especially in peadiatric population, due to anatomical and physiological considerations. If severe or prolonged, this lack of oxygen can result in permanent brain damage, damage to other vital organs or even death. Pre-oxygenation prior to induction of anaesthesia is standard practice to prevent desaturation and hypoxemia. Apnoeic oxygenation in adults is effective and prolongs the time to desaturation. Apneic oxygenation is a novel method of delivering oxygen to a patient despite a lack of active respiration (i.e. the patient is not breathing on their own and the investigators are not providing the patient an artificial breath). The simplest and least invasive method to provide apneic oxygenation is the application of oxygen through nasal cannula during airway management. The effectiveness of apnoeic oxygenation in the adult is well document, especially in bariatric population or ICU, however only few study are interesting about pediatric population. Recent studies suggest that high flow is similar to low flow oxygenotherapy. Therefore, the aim of this study was to investigate the effectiveness of apnoeic oxygenation during airway management in infants.

This is a randomized clinical trial investigating the utility of apneic oxygenation via high flow nasal cannula during airway management for infant's general anesthesia. Three groups will be compared, a control group at 0 L/min, a 0,2L/Kg/min and a 1L/Kg/min group. The primary outcome will be the time (in seconds) between onset of apnea and one of these end-points : desaturation (SPO2 <95%) or Airway management completed.

All infants included will receive french actual standard of care concerning general anesthesia and peri-operative medicine.

ELIGIBILITY:
Inclusion Criteria:

* Infants Between 0 (post-conceptionnal age >41 weeks post Amenorrhea) and 24 months of life
* Scheduled for elective surgery under general anesthesia
* Need of orotracheal Intubation by direct laryngoscopy or Video-laryngoscopy

Exclusion Criteria:

* Emergency surgery
* Crush Induction needed
* High clinical risk of difficult airway management
* Premature before 1 month of life

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-08-04 (Estimated); Study Completion 2020-11-04 (Estimated)

PRIMARY OUTCOMES:
Time between apnoea and issues | Start at the onset of Apnoea
  Time, in seconds, between the onset of Apnoea (No EtCO2 on the capnogram) and one of these two Issues :
  * SpO2< 95%
  * Airway Management Completed (Orotracheal intubation completed and 3 similar capnograms on the respirator)

SECONDARY OUTCOMES:
Minimal SpO2 during the procedure (%) | Between Onset of apnoea and airway management completed
  Minimal SpO2 recorded during the onset of apnoea and airway management completed
Time to SpO2 = 90% (in seconds) | During Airway Management, after Apnoea Onset
  Time between onset of apnoea and SpO2 = 90%, if it occurs, even if mask ventilation is started at Spo2 =95%
Numbers of Laryngoscopy attempts (n) | During Airway management
  Numbers of Laryngoscopy needed to secure Airways
Need to Face Mask Reventilating (Yes/No) | During Airway management
  : Incidence of Face Mask Reventilating during Airway management, needed by Sp02 reach under 95%
Area under SpO2 curve | During Airway management
  AUC of SpO2 recorded every 10 seconds
Respiratory Events (Incidence and type) | During Airway management
  Incidence of respiratory diseases during Airway management (Bronchospasm, Pneumothorax, Laryngospasm, Laryngeal Oedema)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Gerst, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France